CLINICAL TRIAL: NCT00111722
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group, Placebo Controlled Study to Evaluate the Efficacy and Tolerability of Rizatriptan 10 mg Tablets for the Treatment of Menstrual Migraine
Brief Title: Study to Test a Marketed Drug in the Treatment of Menstrual Migraine (0462-072)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0462-072; 2005_025
Record Dates: First submitted 2005-05-24; First posted 2005-05-25 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0462, rizatriptan benzoate / Duration of Treatment -1day
Drug: Comparator: placebo / Duration of Treatment - 1 day

SUMMARY:
The purpose of this study is to test the effectiveness of a marketed drug in the treatment of a menstrual migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Female patient at least 18 years old
* Patient has menses approximately monthly
* Patient has at least a 6 month history of migraine and at least a 6 month history of menstrual migraine

Exclusion Criteria:

* Pregnant and/or nursing mother
* Cardiovascular disease
* Uncontrolled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2005-05-27 (Actual); Primary Completion 2006-02-15 (Actual); Study Completion 2006-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with 2 hour pain relief: 4-point headache severity scale as recorded in patient diary

SECONDARY OUTCOMES:
Percentage of patients with 24-hr sustained pain relief: headache severity between 2 and 24 hrs post dose recorded in patient diary

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Mannix LK, Loder E, Nett R, Mueller L, Rodgers A, Hustad CM, Ramsey KE, Skobieranda F. Rizatriptan for the acute treatment of ICHD-II proposed menstrual migraine: two prospective, randomized, placebo-controlled, double-blind studies. Cephalalgia. 2007 May;27(5):414-21. doi: 10.1111/j.1468-2982.2007.01313.x. PMID 17448179
- [Background] Nett R, Mannix LK, Mueller L, Rodgers A, Hustad CM, Skobieranda F, Ramsey KE. Rizatriptan efficacy in ICHD-II pure menstrual migraine and menstrually related migraine. Headache. 2008 Sep;48(8):1194-201. doi: 10.1111/j.1526-4610.2008.01093.x. Epub 2008 Apr 14. PMID 18422606